CLINICAL TRIAL: NCT03700775
Title: Remote Hypertension Management Using Home Blood Pressure Telemonitoring and a Standardized Treatment Protocol
Brief Title: Hypertension Management Using Telemonitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0012
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Hypertension
Keywords: Hypertension; Telemedicine
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Singe center prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemonitoring intervention (Experimental)
  Interventions: Other: Remote Telemonitoring

INTERVENTIONS:
Other: Remote Telemonitoring — Using the telemedicine kit, participants will record a daily health session including 2 BP measurements obtained one minute apart. Participants are encouraged to record a health session every day, with a minimum of 5 days per week. Participants are also encouraged to equally divide health session recordings between the mornings and evenings. Every 2 weeks BP measurements will be assessed. If less than 75% of measurements are at goal <130/80 mmHg, the central Telehealth pharmacist will designate drug-therapy intensification according to an evidence-based treatment algorithm that is physician approved. Regardless of BP control, participants will be contacted by their nurse coordinator every 2 weeks. During all telephone visits nurse coordinators emphasize healthy lifestyle habits. Safety protocols are in place for dangerously high or low BP recordings.

SUMMARY:
This is a prospective study evaluating the feasibility and safety of remote hypertension management using a central telemonitoring program among patients with elevated blood pressure (BP) at the University of Mississippi Medical Center (UMMC).

DETAILED DESCRIPTION:
Patients with elevated BP, identified by the electronic medical record, will be recruited for study enrollment. Patients will be mailed a telemonitoring kit including an electronic tablet equipped with a wireless BP cuff that transmits measurements directly to the UMMC electronic medical record and monitored by the UMMC Center for Telehealth. Patients will participate in a 6 month intervention period during which they will transmit daily BP recordings with regular contact by a Telehealth nurse coordinator who will provide education and encourage healthy lifestyle habits. Every 2 weeks BP medications will be adjusted according to an evidence-based treatment algorithm managed by the Center for Telehealth pharmacist using a standardized physician-approved protocol. Data analysis will track metrics of study enrollment, study completion, safety, therapeutic intensification, and BP change from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Patient of UMMC clinician approving the study
3. At least 2 clinic encounters in the past 12 months with systolic BP ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg

Exclusion Criteria:

1. Stage 4 or 5 chronic kidney disease
2. Systolic heart failure (LVEF <50%) or major cardiovascular event (MI, stroke) within 3 months
3. Resistant hypertension (prescribed 3 or more antihypertensive medications at target doses) or known secondary cause of hypertension
4. Pregnancy or inability/unwillingness to use birth control for women of child-bearing potential
5. Institutionalized, dementia, limited life expectancy, uncontrolled mental illness, substance abuse, or other conditions that would prohibit ability to perform regular home BP monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Adverse events | 6 months
  Adverse event data will primarily be collected through self-report during each nursing coordinator contact with the patient. Participants will report any hospitalization longer than 12 hours, emergency room visits, or some-day clinic visits and reasons for those visits since the prior nurse coordinator encounter. Study staff will obtain and review medical records related to all adverse events including: deaths, hospitalizations, major cardiac events, incident kidney failure, and urgent evaluations for hypertension, hypotension, loss of consciousness or fainting, allergic reactions, hives, and angioedema. These events are evaluated for severity, expectedness, and potential relatedness to the intervention and study participation.

SECONDARY OUTCOMES:
BP control rates | 12 months
  Number of participants with systolic BP <130 mmHg and diastolic BP <80 mmHg at the first clinic visit following completion of the protocol
Antihypertensive medication adjustments | 6 months
  Quantify dose adjustments of existing medications and initiation of new medications

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
This is a prospective pilot study assessing safety and feasibility.